CLINICAL TRIAL: NCT00398229
Title: The Benefit of Human Chorionic Gonadotropin (hCG) Supplementation Throughout the Secretory Phase of Frozen-Thawed Embryo Transfer Cycles
Brief Title: hCG Supplementation in Frozen-Thawed Embryo Transfer Cycle
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Arik Tzukert, Hadassah Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: freezehcg-HMO-CTIL
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2009-01-01 (Estimated); Status verified 2007-11

CONDITIONS: Fertility Agents, Female
Keywords: In-Vitro Fertilization; human chorionic gonadotropin; frozen-thawed embryo transfer; implantation rate
MeSH Terms: interventions — Chorionic Gonadotropin

ARMS (2):
- A (Active Comparator): receiving hCG injection
  Interventions: Drug: s.c. human chorionic gonadotropin (Ovitrelle)
- B (Placebo Comparator)
  Interventions: Drug: s.c. human chorionic gonadotropin (Ovitrelle)

INTERVENTIONS:
Drug: s.c. human chorionic gonadotropin (Ovitrelle) — S.C. Ovitrelle 250 mcg once

SUMMARY:
The implantation rate after frozen-thawed embryo transfer cycles depends mostly on the receptivity of the endometrium and the embryo quality.The effects of human chorionic gonadotropins (hCG) on the endometrium have been investigated for several years. hCG was shown to up-regulate gene expression during the differentiation of human endometrial stromal cells into decidua. The aim of our study was to assess the benefit of hCG supplementation throughout the secretory phase of artificial frozen-thawed embryo transfer cycles.

ELIGIBILITY:
Inclusion Criteria:

* all women on frozen-thawed embryo-transfer cycle

Exclusion Criteria:

* any allergy to injection of human chorionic gonadotropin before

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-11; Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
implantation rate | 4 weeks
pregnancy rate | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Assaf Ben-Meir, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical center, Jerusalem, Israel